CLINICAL TRIAL: NCT02207959
Title: Endoscopic Multispectral Imaging for the Early Detection of Gastric Neoplasia
Brief Title: Gastric In Vivo Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Susana Gonzalez (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor-Investigator, Susana Gonzalez, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 09-0696B
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Neoplasia; Endoscopic imaging; In vivo imaging
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surveillance Endoscopy (Experimental): White light examination, vital-dye enhanced fluorescence examination (VFI), High Resolution Microendoscope (HRME)
  Interventions: Drug: Proflavine Hemisulphate salt; Procedure: White-light examination; Procedure: Imaging with High Resolution Microendoscope

INTERVENTIONS:
Drug: Proflavine Hemisulphate salt — The stomach will be sprayed with 1-10 ml of 0.01% proflavine using a standard endoscopic spray-catheter.
  Other Names: Vital-dye enhanced fluorescence imaging; VFI
Procedure: White-light examination — standard white light examination
  Other Names: White-light endoscopic examination
Procedure: Imaging with High Resolution Microendoscope — HRME will be inserted through the biopsy channel of the endoscope, gently placed against the mucosa, and images of suspicious areas will be obtained.
  Other Names: HRME; VFI/HRME

SUMMARY:
The overall objective of this pilot study is to determine whether multispectral imaging increases the diagnostic accuracy of the current standard of high-definition white-light endoscopy for the detection of gastric neoplasia (high grade dysplasia or cancer). As part of an NCI-funded RO1, the investigators goal is to develop a multispectral endoscopic platform that can be used to survey a large surface area and, potentially, serve as a "red flag" for microendoscopic imaging of small areas. In prior ex vivo evaluations of surgical and endoscopic specimens, the investigators have identified the optical settings and illumination wavelengths that are complementary to white-light imaging and enhance superficial mucosal and vascular changes associated with neoplasia. Based on this initial testing, vital-dye enhanced fluorescence imaging (VFI) and imaging with High Resolution Microendoscope (HRME) have been identified as modalities that may be complementary to white-light imaging. The goal of this pilot study is to preliminarily determine the accuracy of these modalities during the endoscopic surveillance and detection of gastric neoplasia.

DETAILED DESCRIPTION:
Consent will be obtained the day of the subject's scheduled endoscopy in a clinical room or at a routine office visit prior to the endoscopy. The study investigator will explain the study including the reasons why subject may be eligible, risks, and benefits. The subject will be given a chance to address any questions or concerns they may have.

If the patient agrees to participate in this study all of the procedures listed below will be performed the day of the scheduled endoscopy exam. The procedures listed are part of the routine standard of care for an endoscopy exam, except for the images that are being taken and the additional 2-6 biopsies taken from any abnormal areas that are seen with the new imaging technique. The use of the imaging technique described in this research study will not change the standard of care procedures.

The endoscopic procedure is outlined below:

1. White Light Examination: Examination will initially be performed in the standard white-light endoscopic mode as is routinely done. Abnormal gastric mucosa areas and nodularities will be recorded. Any "Suspicious" areas (visible abnormalities, etc.) will be photographed and the location recorded (distance from incisors and endoscopic quadrant, eq. 34 cm; greater curvature, lesser curvature, etc).
2. Vital-Dye Enhanced Fluorescence Examination: Following this, the stomach will be sprayed with 1-10 ml of 0.01% proflavine using a standard endoscopic spray-catheter. Using the fluorescent imaging, the location of any VFI-"Suspicious' areas will be recorded. Additionally, VFI examination of any suspicious areas seen on WLE will be performed. The endoscopist will label the surface-appearance of each WLE abnormal area based on its VFI appearance. Thus, each area will be labeled as: "Not Suspicious," or "Suspicious for Neoplasia."
3. HRME examination: WLE and VFI suspicious appearing areas will be further imaged with HRME. HRME will be inserted through the biopsy channel of the endoscope, gently placed against the mucosa, and images of suspicious areas will be obtained. The endoscopist will label the surface-appearance of each WLE abnormal area and VFI abnormal area, based on the HRME appearance. Thus, each area will be labeled as: "Not Suspicious," or "Suspicious for Neoplasia."
4. Biopsy Protocol: Biopsies will be obtained of any area suspicious on any of the imaging modalities (WLE, VFI or HRME). Additionally, two 'control' areas (normal on imaging) will also be biopsied. Lastly, routine, biopsies will be performed per clinical care to determine areas of intestinal metaplasia and H pylori infection as per routine standard of care.
5. Pathologic Interpretation: All samples will be evaluated by a single expert gastrointestinal pathologist who will be blinded to the endoscopic findings

ELIGIBILITY:
Inclusion Criteria:

* patients with high grade dysplasia in the stomach and known or suspected cancer of the stomach undergoing endoscopic surveillance
* at least 18 years of age

Exclusion Criteria:

* subjects who report an allergy to Proflavine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Gastric neoplasia presence | Day 1
  Comparison of the efficiency of widefield imaging modality or combination of modalities (WLE, WLE+VFI/HRME for the highest accuracy on the detection of gastric neoplasia

SECONDARY OUTCOMES:
Sensitivity for the detection of neoplasia | Day 1
  the potential errors in estimation of sensitivity (true positive rate)
Specificity for the detection of neoplasia | Day 1
  the potential errors in estimation of specificity (true negative rate)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Gonzalez, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States